CLINICAL TRIAL: NCT01521702
Title: Adjuvant Gemcitabine Versus NEOadjuvant Gemcitabine/Oxaliplatin Plus Adjuvant Gemcitabine in Resectable PAncreatic Cancer: a Randomized Multicenter Phase III Study
Brief Title: NEOadjuvant Gemcitabine/Oxaliplatin Plus Adjuvant Gemcitabine in Resectable PAncreatic Cancer
Acronym: NEOPAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOPAC / IPC 2011-002
Record Dates: First submitted 2011-12-22; First posted 2012-01-31 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Pancreas Cancer
Keywords: adenocarcinoma; pancreatic head
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Neoadjuvant Therapy; Surgical Procedures, Operative; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neoadjuvant chemotherapy (Experimental): After initial staging laparoscopy, Neoadjuvant chemotherapy consists of four bi-weekly cycles of gemcitabine (intravenous infusion of 1000mg/m2 over 30 minutes) and oxaliplatin (intravenous infusion of 100mg/m2 over 2 hours, modified from the Louvet protocol11).
  Interventions: Drug: Neoadjuvant chemotherapy
- surgery (Active Comparator): surgery
  Interventions: Procedure: surgery and Adjuvant chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — four bi-weekly cycles of gemcitabine (intravenous infusion of 1000mg/m2 over 30 minutes) and oxaliplatin (intravenous infusion of 100mg/m2 over 2 hours,
  Arms: Neoadjuvant chemotherapy
Procedure: surgery and Adjuvant chemotherapy — surgery and Adjuvant chemotherapy must be started within eight weeks after surgery and is based on the standard regimen using six cycles of gemcitabine (Gem 1000mg/m2 over 30 minutes) on days 1, 8, 15 every 4 weeks.
  Arms: surgery

SUMMARY:
The aim of this study is to test the additional value of neoadjuvant chemotherapy to the standard treatment for resectable pancreatic cancer (surgery + adjuvant chemotherapy).

This study will be performed in compliance with the study protocol, GCP (good clinical practice) and the applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* resectable adenocarcinoma of the pancreatic head (requiring duodeno-pancreatectomy)
* T1-3, Nx, M0 (UICC 6th version, 2002)
* infiltration of the portal vein (<180°) is not an exclusion criterion
* cytologic or histologic confirmation of adenocarcinoma
* age >18 years
* written informed consent

Exclusion Criteria:

* contraindication for Whipple procedure
* an infiltration >180° of the portal vein
* abutment of the tumor to the superior mesenteric artery
* infiltration of the superior mesenteric artery or the celiac trunk
* chronic neuropathy > grade 2
* WHO performance score >2
* uncorrectable cholestasis (bilirubin > 100mmol/l despite drainage attempts for more than four weeks prior to inclusion)
* female patients in child bearing age not using adequate contraception (oral or subcutaneous contraceptives, intrauterine pessars (IUP), condoms)
* pregnant or lactating women
* mental or organic disorders which could interfere with giving informed consent or receiving treatments
* Second malignancy diagnosed within the past 5 years, except non-melanomatous skin cancer or non-invasive cervical cancer
* percutaneous biopsy of the primary tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
progression-free survival | from date of randomization until date of progression, assessed up to 5 years
  period from study inclusion until the date of recurrence or surgery (in case of unresectability at surgical exploration).

SECONDARY OUTCOMES:
histology | at 6 months
  histological response,
overall survival | From date of randomization until date of death, assessed up to 5 years
  time from date of inclusion to date of death
complication | until 6 months
  complication rates after surgery,

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc RAOUL, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr